CLINICAL TRIAL: NCT03715803
Title: Calistar A vs. Calistar S - Cohort Retrospective Analysis
Brief Title: Calistar A vs. Calistar S - Comparative Cohort Retrospective Analysis of Single Incision POP Systems
Status: Completed | Type: Observational
Sponsor: Agustin Sampietro (Other)
Responsible Party: Sponsor-Investigator, Agustin Sampietro, Gynecologist, University of Buenos Aires
Organization: University of Buenos Aires (Other)
Other Study IDs: CaSCaA
Record Dates: First submitted 2018-09-26; First posted 2018-10-23 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calistar A: Calistar A mesh to treat anterior and apical POP
  Interventions: Device: Calistar A mesh to treat anterior and apical POP
- Calistar S: Calistar S mesh to treat anterior and apical POP
  Interventions: Device: Calistar S mesh to treat anterior and apical POP

INTERVENTIONS:
Device: Calistar A mesh to treat anterior and apical POP — Single incision surgery using Calistar A mesh to treat anterior and apical pelvic prolapses
  Groups: Calistar A
Device: Calistar S mesh to treat anterior and apical POP — Single incision surgery using Calistar S to treat anterior and apical pelvic prolapses
  Groups: Calistar S

SUMMARY:
The main objective of this study is to compare the initial outcomes and complication of two meshes implanted through a single incision to treat anterior and apical prolapses, Calistar A and a second-generation low weight mesh called Calistar S (Soft).

DETAILED DESCRIPTION:
The main objective of this study is to compare the initial outcomes and complication of two meshes implanted through a single incision to treat anterior and apical prolapses, Calistar A and a second-generation low weight mesh called Calistar S (Soft). In such sense, objective and subjective parameters will be retrospectively tested to demonstrate the safety and effectiveness of this products. Safety will be assessed by register of complications and effectiveness will be evaluated by pelvic floor reconstruction and quality of life improvements.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Anterior and apical prolapse Stage 3 (according to POP-Q) or more with or without stress urinary incontinence (SUI)
* Primary or recurrent treatment with Calistar S or Calistar A
* At least 6 months follow-up

Exclusion Criteria:

* Recurrent vaginal infections,
* Chronic colorectal diseases (chronic nonspecific ulcerative colitis, diverticulitis, diverticulosis, Chron's disease, irritable bowel syndrome, familial polyposis).
* Presence of any coagulopathies,
* Impairment of the immune system or any condition that compromises recovery,
* Prior irradiation
* Chronic pelvic pain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults female
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustín Sampietro, Dr, Principal Investigator — Faculty of Medicine, University of Buenos Aires
Locations (1):
- Hospital Británico, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
Only final clinical study report will be shared with the researchers participating in the study

REFERENCES:
- [Background] de Tayrac R, Madelenat P. [Evolution of surgical routes in female stress urinary incontinence]. Gynecol Obstet Fertil. 2004 Dec;32(12):1031-8. doi: 10.1016/j.gyobfe.2004.10.019. French. PMID 15589779
- [Background] Bigozzi MA, Provenzano S, Maeda F, Palma P, Riccetto C. In vivo biomechanical properties of heavy versus light weight monofilament polypropylene meshes. Does the knitting pattern matter? Neurourol Urodyn. 2017 Jan;36(1):73-79. doi: 10.1002/nau.22890. Epub 2015 Oct 5. PMID 26436858
- [Background] Barber MD, Brubaker L, Nygaard I, Wheeler TL 2nd, Schaffer J, Chen Z, Spino C; Pelvic Floor Disorders Network. Defining success after surgery for pelvic organ prolapse. Obstet Gynecol. 2009 Sep;114(3):600-609. doi: 10.1097/AOG.0b013e3181b2b1ae. PMID 19701041
- [Background] Toozs-Hobson P, Freeman R, Barber M, Maher C, Haylen B, Athanasiou S, Swift S, Whitmore K, Ghoniem G, de Ridder D; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for reporting outcomes of surgical procedures for pelvic organ prolapse. Neurourol Urodyn. 2012 Apr;31(4):415-21. doi: 10.1002/nau.22238. PMID 22517068
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calistar A | Calistar S
Started | 91 | 126
Completed | 91 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calistar A | Calistar S | Total
Number analyzed (Participants) | 91 | 126 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 62 (8) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 126 | 217
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 32 | 71 | 103
  Brazil | 23 | 19 | 42
  Italy | 29 | 30 | 59
  France | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cured Participants According to Barber Criteria
Description: According to Barber criteria cure is defined if there are no points beyond the hymen (measure by POP-Q quantification), an absence of vaginal bulge symptoms and no re-treatment/interventions on year post procedure.
Time Frame: Post-operative at 6 months
Measure: Number; unit: percentage of cured patients
Arm/Group | Calistar A | Calistar S
Number analyzed (Participants) | 91 | 126
percentage of cured patients | 82.42 | 90.48

2. Secondary Outcome: Percentage of Participants Cured According to Objective Measure (POP-Q Quantification)
Description: Assessment of POP with POP-Q quantification. Number of participants cured according to POP-Q quantification. Success criteria: POP-Q stage equal 0 or 1.
Time Frame: Pre-operative and post-operative at 6 months
Measure: Number; unit: percentage of cured patients
Arm/Group | Calistar A | Calistar S
Number analyzed (Participants) | 91 | 126
percentage of cured patients | 82.42 | 88.88

3. Secondary Outcome: Quality of Life Status: Patient Global Impression Questionnaire
Description: Patient satisfaction with the experience and the result of procedure will be evaluated with the "Patient Global Impression" questionnaire. This is a visual analogue scale range 1 (very much worse) - 5 (very much improved). A higher score a better outcome.
Time Frame: Post-operative at 6 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Calistar A | Calistar S
Number analyzed (Participants) | 91 | 126
units on a scale | 5 [1 to 5] | 5 [3 to 5]

4. Secondary Outcome: Adverse Events
Description: Register of adverse events. Clavien-Dindo classification
Time Frame: Intra-operative and post-operative at 6 months
Population: Adverse events were presented in a separate section.
Arm/Group | Calistar A | Calistar S
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Quality of Life: PFDI 20
Description: Quality of life assessed with "Pelvic Floor Distress Inventory (PFDI 20)" questionnaire to evaluate the impact of urinary, prolapse and colorectal distress post-operative. The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 (least distress) to 100 (greatest distress).
Time Frame: Post-operative at 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Calistar A | Calistar S
Number analyzed (Participants) | 91 | 126
score on a scale | 30.85 [0 to 91.1] | 19.4 [0 to 52.8]

6. Other Pre Specified Outcome: Quality of Life: PISQ-12
Description: Quality of life assessed with "Pelvic Organ Prolapse/ Urinary Incontinence Sexual Questionnaire (PISQ-12)" to evaluate sexual function in women with pelvic organ prolapse and/or urinary incontinence post-operative. Higher PISQ-12 scores indicate a better sexual function. Maximum score is 48.
Time Frame: Post-operative at 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Calistar A | Calistar S
Number analyzed (Participants) | 91 | 126
score on a scale | 0 [0 to 5] | 0 [0 to 13]

ADVERSE EVENTS:
Time Frame: All adverse events were collected within a FU of 24 mo (6-64 mo) for Ca A and 12 mo (6-36 mo) for Ca S
Arm/Group | Calistar A | Calistar S
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/126
Other Adverse Events (participants affected / at risk) | 30/91 | 14/126
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calistar A (N=91) | Calistar S (N=126)
Pain (Surgical and medical procedures) | 6 (6) | 6 (6)
Reoperation for prolapse (Surgical and medical procedures) | 2 (2) | 2 (2)
Mesh erosion (Surgical and medical procedures) | 10 (10) | 5 (5)
Urinary tract infection (Renal and urinary disorders) | 12 (12) | 1 (1)

LIMITATIONS AND CAVEATS:
Retrospective study; CaA procedures started a long time before the first CaS cases (Ca S level of surgeon training more experienced). Available data only enables mid-term follow-ups of differing duration's between the two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03715803/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03715803/SAP_001.pdf